CLINICAL TRIAL: NCT00543127
Title: Phase III Trial Comparing Efficacy and Tolerance of Fulvestrant for 3 Years (y) Combined With Anastrozole 5 y Versus Anastrozole 5 y as Adjuvant Hormonotherapy in Postmenopausal With Early Breast Cancer and Positive Hormone Receptors
Brief Title: Fulvestrant (Faslodex) + Anastrozole (Arimidex) vs Anastrozole
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unjustified decision of company that funded the trial.
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2006-10; 2007-003417-14 (EudraCT Number)
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: luminal; anastrozole; fulvestrant; early breast cancer; HR+/HER2-
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fulvestrant + Anastrozole (Experimental): Fulvestrant loading dose regimen will consist of two 5 ml intramuscular injections on day 0 (500 mg), 250 mg single injection on days 14 and 28, and 250 mg single injection every 28 days thereafter for 3 years plus Anastrozole 1 mg PO once daily for 5 years
  Interventions: Drug: Fulvestrant; Drug: Anastrozole
- Anastrozole (Active Comparator): Anastrozole 1 mg will be administered orally as one tablet daily for 5 years.
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Fulvestrant — 500 mg Im Fulvestrant day 0, 250 mg days 14 and 28(charge dose); later 250 mg each 28 days during 3 years plus 1 mg oral Anastrozole per day during 5 years.
  Other Names: Faslodex
  Arms: Fulvestrant + Anastrozole
Drug: Anastrozole — 1 mg oral Anastrozole per day during 5 years.
  Other Names: Arimidex

SUMMARY:
Postmenopausal women with hormone receptor positive and negative Her2 tumours.

Before randomization, the patients will be stratified according to the center, positive nodes (0 vs. 1-3 vs. ≥4), previous chemotherapy (yes vs no) and hormonal receptors status.

DETAILED DESCRIPTION:
It is expected that disease-free survival for patients receiving Anastrozole alone for 5 years will be up to 90%. An increase of 3% in disease-free survival (DFS) is expected in the arm of Fulvestrant plus Anastrozole, i.e a DFS of up to 93%. They will be required 1358 patients per treatment group (i.e, 2716 patients in total) to give 80% power, alfa bilateral 0.05, and OR 0.6888. Assuming 5% screening failures 2852 patients are required to enter the study. In Jun-2010 the recruitment was stopped due to lack of support of the financier based on the result of Faslodex® and Arimidex® in Combination Trial (FACT-trial), comparing Fulvestrant + Anastrozole vs Anastrozole alone in 1st relapse showed no difference in time to progression at more than 40 months follow-up.

ELIGIBILITY:
Inclusion criteria:

1. Histological documentation of breast cancer.
2. Stage I, II, IIIA and IIIC* invasive breast cancer. One of these two characteristics must be fulfilled:

   * N+
   * T > 1cm *Eligible patients T1-T3 and pN3a (patients with metastasis in infraclavicular nodes would not be eligible)
3. Local treatment with curative intention:

   * mastectomy or tumour excision with free margins + radiotherapy
   * axillary lymphadenectomy or sentinel node biopsy
4. Positive hormone receptors (Estrogen Receptor [ER]+ and/or Progesterone Receptor [PR]+) in primary tumour tissue as measured by a central laboratory
5. Human Epidermal Growth Factor Receptor 2 (HER2) negative breast cancer, defined as immunohistochemistry (IHC) 0 or 1+ or negative fluorescence in situ hybridization (FISH) (in the event of IHC 2+ or 3+)
6. Postmenopausal women, defined as women meeting any of the following criteria:

   * Age ≥ 60 years
   * Age ≥ 45 years with amenorrhea ≥ 12 months in the moment of breast cancer diagnosis and an intact uterus
   * Prior bilateral ovariectomy
   * In case previous hysterectomy, follicle stimulating hormone (FSH) and estradiol levels within the postmenopausal range (using local laboratory ranges)* * In patients previously treated with a luteinizing hormone releasing hormone (LH-RH) analogue, the last extended release formulation should have been administered more than 6 months before randomisation, and menses must not have reappeared.
7. A World Health Organization (WHO) performance status of 0, 1, or 2.
8. Age > 18 years

Exclusion criteria:

1. Presence of metastatic disease or bilateral invasive cancer
2. ER and Progesterone Receptor (PR) negative breast cancer
3. HER2-positive breast cancer, defined as FISH+
4. Treatment with a non-approved or experimental drug within 4 months of randomisation
5. Current malignancy or previous malignancy in the past 5 years (other that breast cancer or basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix)
6. Pregnant or nursing patients
7. Any of the following laboratory values within 3 months of randomisation:

   * Platelets < 100 x 109/L
   * Total bilirubin > 1.5 x Upper limit of reference range (ULRR)**

     ** Patients with documented Gilbert syndrome may be included in this trial
   * Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) > 2.5 x ULRR
   * A history of:
   * hemorrhagic diathesis (i.e. Disseminated Intravascular Coagulation [DIC], coagulation factor deficiency) or
   * long-term anticoagulant treatment (except for anti-platelet aggregants and low-dose warfarin; see section 3.7)
8. A history of hypersensitivity to the active ingredient or inactive excipients of fulvestrant, aromatase inhibitors, or castor oil
9. Any concomitant severe disease advising against patient participation in the trial o that may jeopardize compliance with the trial protocol, such as uncontrolled heart disease, uncontrolled diabetes mellitus, or uncontrolled severe infections
10. Hormone replacement therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital General Universitario Gregorio Marañón; Study Director, Study Director — Centro Oncológico de Galicia; Study Director, Study Director — Hospitales Universitarios Virgen del Rocío
Locations (53):
- Spain (53):
  - Hospital Universitario Virgen de Los Lirios, Alcoy, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital General Universitario de Elda, Elda, Alicante
  - Hospital Usp San Jaime, Torrevieja, Alicante
  - Hospital de Torrevieja Salud Ute, Torrevieja, Alicante
  - Hospital Municipal de Badalona, Badalona, Barcelona
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Institut Catalá D'Oncología L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castellón
  - Hospital Donostia, Donostia / San Sebastian, Guipúzcoa
  - Onkologikoa, Donostia / San Sebastian, Guipúzcoa
  - Hospital de Barbastro, Barbastro, Huesca
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital San Agustín de Avilés, Avilés, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa CRUZ DE Tenerife
  - Hospital Universitario de Valme, Dos Hermanas, Sevilla
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Lluís Alcanyis, Xátiva, Valencia
  - Hospital de Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Centro Oncológico de Galicia, A Coruña
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - HOSPITAL UNIVERSITARI DE GIRONA DR. JOSEP TRUETA (ICO de Girona), Girona
  - Hospital Universitario San Cecilio, Granada
  - Hospital General Universitario de Guadalajara, Guadalajara
  - Hospital Juan Ramón Jiménez, Huelva
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - CENTRO INTEGRAL ONCOLÓGICO CLARA CAMPAL (Hospital Madrid Norte Sanchinarro), Madrid
  - Hospital Clínico Universitario Virgen de La Victoria, Málaga
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Del Rocío, Seville
  - Hospital Virgen de La Salud, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Arnau de Vilanova de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Result] Ruiz-Borrego M, Guerrero-Zotano A, Bermejo B, Ramos M, Cruz J, Baena-Canada JM, Cirauqui B, Rodriguez-Lescure A, Alba E, Martinez-Janez N, Munoz M, Antolin S, Alvarez I, Del Barco S, Sevillano E, Chacon JI, Anton A, Escudero MJ, Ruiz V, Carrasco E, Martin M; GEICAM. Phase III evaluating the addition of fulvestrant (F) to anastrozole (A) as adjuvant therapy in postmenopausal women with hormone receptor-positive HER2-negative (HR+/HER2-) early breast cancer (EBC): results from the GEICAM/2006-10 study. Breast Cancer Res Treat. 2019 Aug;177(1):115-125. doi: 10.1007/s10549-019-05296-8. Epub 2019 May 31. PMID 31152327
- [Derived] Martin M, Carrasco E, Rodriguez-Lescure A, Andres R, Servitja S, Anton A, Ruiz-Borrego M, Bermejo B, Guerrero A, Ramos M, Santaballa A, Munoz M, Cruz J, Lopez-Tarruella S, Chacon JI, Alvarez I, Martinez P, Miralles JJ, Polonio O, Jara C, Aguiar-Bujanda D. Long-term outcomes of high-risk HR-positive and HER2-negative early breast cancer patients from GEICAM adjuvant studies and El Alamo IV registry. Breast Cancer Res Treat. 2023 Sep;201(2):151-159. doi: 10.1007/s10549-023-07002-1. Epub 2023 Jun 20. PMID 37338729
- See also: Description Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 870 patients were recruited, from them, 437 were randomized to Anastrozole (A) and 433 to A plus Fulvestrant (F), but 18 patients (3 in A arm and 15 in arm A+F) never received treatment.
Groups:
- Fulvestrant + Anastrozole: Fulvestrant + Anastrozole: 500 mg Im Fulvestrant day 0, 250 mg days 14 and 28(charge dose); later 250 mg each 28 days during 3 years plus 1 mg oral Anastrozole per day during 5 years.
Period: Overall Study
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Started | 433 | 437
Completed | 303 | 350
Not Completed | 130 | 87

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant + Anastrozole | Anastrozole | Total
Number analyzed (Participants) | 433 | 437 | 870
Age, Continuous [Median (Full Range); unit: years] | 62 [40 to 86] | 62 [44 to 86] | 62 [40 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 433 | 437 | 870
  Male | 0 | 0 | 0
Breast Surgery [Count of Participants; unit: Participants]
  Conservative | 303 | 310 | 613
  Mastectomy | 130 | 127 | 257
Axillary surgery [Count of Participants; unit: Participants]
  Axillary dissection | 258 | 281 | 539
  Sentinel Node Biopsy | 174 | 155 | 329
  Unknown | 1 | 1 | 2
Previous chemotherapy [Count of Participants; unit: Participants]
  Adjuvant | 256 | 261 | 517
  Neoadjuvant | 37 | 34 | 71
  Neoadjuvant + Adjuvant | 3 | 2 | 5
  None | 137 | 140 | 277
Previous radiotherapy [Count of Participants; unit: Participants]
  YES | 348 | 347 | 695
  NO | 85 | 90 | 175
Histopathologic type [Count of Participants; unit: Participants]
  Invasive Ductal Carcinoma | 337 | 346 | 683
  Invasive Lobular Carcinoma | 71 | 71 | 142
  Other | 25 | 20 | 45
Histologic grade [Count of Participants; unit: Participants] — The grade of a breast cancer is a prognostic factor and is representative of the "aggressive potential" of the tumor. In a broad generalization, "low grade" cancers tend to be less aggressive than "high grade" cancers. There are 3 grades: Grade I tumors have a total score of 3-5, Grade II tumors have a total score of 6-7 and Grade III tumors have a total score of 8-9. Grade X is unknown result.
  Participants
    Grade 1 | 88 | 82 | 170
    Grade 2 | 216 | 235 | 451
    Grade 3 | 94 | 83 | 177
    Grade X | 35 | 37 | 72
Tumor size [Median (Full Range); unit: cm] | 2 [0.08 to 10] | 2 [0.0 to 15] | 2 [0.0 to 15]
Final diagnosis tumor size [Count of Participants; unit: Participants] — Using the Tumour Node Metastasis staging system (TNM) after surgery, the "T" plus a number (0 to 4) is used to describe the size of the tumor. The T0 means the lower size, and the T4 means the higher size. TX means unknown.
  Participants
    T1 | 220 | 243 | 463
    T2 | 189 | 179 | 368
    T3-T4 | 22 | 14 | 36
    TX | 2 | 1 | 3
Nodal status [Count of Participants; unit: Participants] — The "N" in the TNM staging stands for lymph nodes. NX: not evaluated. N0: No cancer was found / Only areas of cancer smaller than 0.2 mm. N1: The cancer has spread to 1 to 3 axillary lymph nodes and/or the internal mammary lymph nodes. N2: The cancer has spread to 4 to 9 axillary lymph nodes, or it has spread to the internal mammary lymph nodes, but not the axillary lymph nodes. N3: The cancer has spread to 10 or more axillary lymph nodes, or it has spread to the lymph nodes located under the clavicle, or collarbone. It may have also spread to the internal mammary lymph nodes.
  Participants
    N0 | 214 | 200 | 414
    N1 | 157 | 164 | 321
    N2 | 42 | 52 | 94
    N3 | 14 | 18 | 32
    NX | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS) Events
Description: Disease-free survival (DFS) has been evaluated in patients treated with Fulvestrant for 3 years and Anastrozole for 5 years as compared to DFS in patients treated with anastrozole for 5 years.
  DFS event is defined as the evidence of local and/or distant recurrence, new primary breast tumour, or death from any cause.
Time Frame: Up to 5 years
Population: Primary statistical analyses of the efficacy outcome variables will be based on an intent-to-treat (ITT) method and will include all randomised patients
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 433 | 437
Participants | 49 | 62

2. Secondary Outcome: Breast Cancer Specific Survival (BCsS) Events
Description: BCsS events has been evaluated in patients treated with Fulvestrant for 3 years and Anastrozole for 5 years as compared to BCsS in patients treated with anastrozole for 5 years.
  BCsS event is defined as the death from breast cancer.
Time Frame: Up to 5 years
Population: Analyses of the efficacy outcome variables will be based on an intent-to-treat (ITT) method and will include all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 433 | 437
Participants | 17 | 18

3. Secondary Outcome: Overall Survival (OS) Event
Description: OS event has been evaluated in patients treated with Fulvestrant for 3 years and Anastrozole for 5 years as compared to DFS in patients treated with anastrozole for 5 years.
  OS event is defined as the death from any cause.
Time Frame: Up to 5 years
Population: Statistical analyses of the efficacy outcome variables will be based on an intent-to-treat (ITT) method and will include all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 433 | 437
Participants | 28 | 34

4. Secondary Outcome: Time to Recurrence (TR) Event
Description: TR event has been evaluated in patients treated with Fulvestrant for 3 years and Anastrozole for 5 years as compared to DFS in patients treated with anastrozole for 5 years.
  TR event is defined as the evidence of breast cancer recurrence (local and/or distant recurrence of breast cancer, does not include second primary malignancies or deaths from any cause).
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Number analyzed (Participants) | 433 | 437
Participants | 36 | 46

ADVERSE EVENTS:
Time Frame: Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs) will be recorded from the date informed consent is signed, during the treatment period, and for up to 8 weeks after the last injection in patients randomised to fulvestrant if this patient does not continue with anastrozole, or up to 30 days after the last tablet when this is the last study treatment received by the patient.
Description: These Adverse Events are by patient (not per cycle). Only grades 2, 3 and 4 are specified.
Arm/Group | Fulvestrant + Anastrozole | Anastrozole
Serious Adverse Events (participants affected / at risk) | 40/415 | 61/437
Other Adverse Events (participants affected / at risk) | 192/415 | 197/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant + Anastrozole (N=415) | Anastrozole (N=437)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
chronic lymphocytic leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
lymphoblastic leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Conduction abnormality/atrioventricular heart block - av block-second degree mobitz type ii (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia - atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia - sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 2 (2) | 1 (1)
Angor (Cardiac disorders) | 0 (0) | 1 (1)
dilated cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Valvular heart disease (Cardiac disorders) | 0 (0) | 2 (2)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
melanoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
t-cell lymphoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
goitre (Endocrine disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Gastritis (including bile reflux gastritis)
Ileus, gi (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colon cancer (Gastrointestinal disorders) | 3 (3) | 3 (3)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectum cancer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Transverse colon adenocarcinoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perforation, gi - appendix (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ulcer, gi - duodenum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhage, CNS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage, gi - colon (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhage, gi - stomach (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 (0) | 1 (1)
acute hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
cholelithiasis (Hepatobiliary disorders) | 1 (1) | 3 (3)
pancreas cancer (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pancreatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutrophils (anc <1.0 x 109 (Infections and infestations) | 0 (0) | 1 (1) — pulmonary/upper respiratory - lung (pneumonia)
Infection with normal ANC or grade 1 or 2 neutrophils dermatology/skin skin (cellulitis) (Infections and infestations) | 1 (1) | 1 (1)
Infection with normal ANC or grade 1 or 2 neutrophils - pulmonary/upper respiratory bronchus (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or grade 1 or 2 neutrophils - pulmonary/upper respiratory lung (pneumonia) (Infections and infestations) | 3 (3) | 0 (0)
Infection with normal ANC or grade 1 or 2 neutrophils - pulmonary/upper respiratory upper airway nos (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or grade 1 or 2 neutrophils - sexual/reproductive function vagina and vulv (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC - cardiovascular heart (endocarditis) (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC - gastrointestinal appendix (Infections and infestations) | 1 (1) | 1 (1)
Infection with unknown ANC - gastrointestinal dental-tooth (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC - pulmonary/upper respiratory lung (pneumonia) (Infections and infestations) | 1 (1) | 2 (2)
Infection with unknown ANC - renal/genitourinary urinary tract nos (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Other: tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 4 (4)
Neuropathy: craneal - cn vi downward, inward movement of eye (Nervous system disorders) | 0 (0) | 1 (1)
glioblastoma multiforme (Nervous system disorders) | 1 (1) | 0 (0)
Meningioma (Nervous system disorders) | 0 (0) | 1 (1)
Traffic accident (Social circumstances) | 0 (0) | 1 (1)
Gastrointestinal abdomen nos pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Musculoskeletal back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pulmonary/upper respiratory chest/thorax nos pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cystocele (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Secondary malignancy - possiby related to cancer treatment, specify: kidney cancer (Renal and urinary disorders) | 1 (1) | 0 (0)
Secondary malignancy - possiby related to cancer treatment, specify: uterine cervix cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast nodule (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Microcalcification in breast (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Flu-like syndrome (General disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 3 (3)
Gastric difuse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infection with normal ANC or grade 1 or 2 neutrophils - renal/genitourinary kidney (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or grade 1 or 2 neutrophils - renal/genitourinary urinary tract nos (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant + Anastrozole (N=415) | Anastrozole (N=437)
Hypertension (Cardiac disorders) | 41 (41) | 58 (58)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 49 (49) | 23 (23)
Weight gain (General disorders) | 39 (39) | 31 (31)
Weight loss (General disorders) | 37 (37) | 41 (41)
Hot flashes/flushes (Endocrine disorders) | 23 (23) | 18 (18)
Cholesterol, serum-high (hypercholesterolemia) (Metabolism and nutrition disorders) | 21 (21) | 23 (23)
LDL-cholesterol high (Metabolism and nutrition disorders) | 22 (22) | 41 (41)
Musculoskeletal bone pain (Musculoskeletal and connective tissue disorders) | 39 (39) | 34 (34)
Musculoskeletal joint pain (Musculoskeletal and connective tissue disorders) | 83 (83) | 81 (81)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No